CLINICAL TRIAL: NCT03484364
Title: Engaging Native Hawaiian/Pacific Islanders and Activating Communities to Take Steps (ENACTS)
Acronym: ENACTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Responsible Party: Principal Investigator, Denise Dillard, Professor, Washington State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U54MD011240 127687; U54MD011240 (NIH)
Record Dates: First submitted 2018-03-15; First posted 2018-03-30 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The ENACTS intervention is four peer-facilitated educational classes delivered over 8 weeks focused on hypertension self-management.
  Interventions: Behavioral: ENACTS
- Waitlist Group (No Intervention): Usual care and $50 in groceries every other week for 8 weeks.

INTERVENTIONS:
Behavioral: ENACTS — Peer-facilitated, self-care BP education delivered every other week for 8 weeks emphasizing healthy diet, traditional NHPI foods, adherence to medication, and encouragement to increase physical activity and stop smoking, with text messaging to boost adherence. $50 of groceries every other week (4 times) over 8 weeks.
  Other Names: Healthy Hearts Among Pacific Islanders (HHAPI)
  Arms: Intervention Group

SUMMARY:
Our Specific Aims are:

1. At the individual level, to compare within-person change in BP and secondary outcomes between the intervention and control groups.
2. At the family level, to evaluate ENACTS' effects on BP and secondary outcomes as within-person change in family members who provide primary support, and as mean change in other adult family members who are not directly engaged in the intervention.
3. At the policy level, to evaluate the intervention's ability to influence grocery store policy on clearly identifying foods that are low in sodium or high in potassium, some of which might not be easily identified with existing labels (e.g., fresh produce). ENACTS combines empirically supported elements of existing programs, thus increasing its probability of success. It aligns with the American Heart Association's call for multilevel prevention.

DETAILED DESCRIPTION:
This study adapts an existing educational intervention to address self-management of hypertension in NHPIs. The multilevel 6-month intervention - "Engaging NHPIs and Activating Communities to Take Steps" (ENACTS) - will use peer-facilitated, self-care BP education delivered weekly for 8 weeks emphasizing healthy diet, traditional NHPI foods, adherence to medication, and encouragement to increase physical activity and stop smoking; with text messaging to boost adherence. ENACTS will be implemented as a randomized controlled trial at 3 community sites serving NHPIs in the Puget Sound area of Washington. 270 NHPI adults (90 per site) with a self-reported physician diagnosis of hypertension and elevated BP measured at enrollment will be randomized to either ENACTS or usual care.

The primary outcome is change in systolic BP. Secondary outcomes are food purchasing behaviors (online ordering, grocery receipts); medication adherence; social support; smoking cessation; and GIS data on daily energy expenditure. The study will use a Geographic Information Systems (GIS) mobile phone app to track participants. Outcomes will be measured at baseline, weekly, at 8 weeks, and at 6 months. The study will also examine change in household food purchasing patterns, enhanced family support for BP control, and BP improvement among family members. A subset of intervention participants and family members will be invited to participate in a program that uses personal photographs for narrative art projects to promote labeling of healthy foods by local retail outlets.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported physician diagnosis of hypertension and/or type 2 diabetes confirmed by a prescription for an anti-hypertensive medication and/or type 2 diabetes medication;
* Self-reported NHPI race;
* *Age 18 years and older at enrollment;
* Measured systolic BP ≥ 140 mmHg on enrollment; measured baseline fasting glucose >125
* reliable internet access
* computer or Smartphone
* current email address
* *Ability to understand written and spoken English; and
* *Ability and willingness to follow all study protocols.

Exclusion Criteria:

* Pregnant or planning on becoming pregnant throughout the course of the study;
* Currently undergoing dialysis or treatment for a terminal illness;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure | 6 months
  Automatic blood pressure

SECONDARY OUTCOMES:
Eating Behaviors | 6 months
  24 hour dietary recall
Food Purchasing | 6 months
  Grocery receipts
Medication Adherence | 6 months
  Hill Bone High Blood Pressure Compliance Scale
Social Support | 6 months
  Family care climate questionnaire
Tobacco Use | 6 months
  National Health Interview Survey
Daily Energy Expenditure | 6 months
  International Physical Activity Questionnaire (IPAQ)

CONTACTS AND LOCATIONS:
Overall Officials: denise dillard, Principal Investigator — Washington State University
Locations (1):
- National Recruitment via Facebook and Internet, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No